CLINICAL TRIAL: NCT03859505
Title: Effects of Photobiomodulation Therapy on Inflammatory Mediators in Patients With Chronic Non-specific Low Back Pain: a Randomized Placebo-controlled Trial
Brief Title: Photobiomodulation Therapy on Inflammatory Mediators on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); University of Bergen (Other)
Responsible Party: Principal Investigator, Shaiane da Silva Tomazoni, Postdoctoral fellow and visiting researcher, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/1361
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Photobiomodulation Therapy; PBMT; Low-Level Laser Therapy; LLLT
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The mode of intervention (active or placebo PBMT) will be coded by an independent researcher. The randomization schedule will contain only codes (not the actual intervention). The output from the PBMT device is exactly the same from either the active or the placebo interventions. These features will guarantee that participants, therapists and outcomes assessor will be blinded to the treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo PBMT (Placebo Comparator): Application of PBMT (Photobiomodulation Therapy) without any dose (0 Joule).
  Interventions: Device: Placebo PBMT
- Active PBMT (Active Comparator): Application of PBMT (Photobiomodulation Therapy) active.
  Interventions: Device: Active PBMT

INTERVENTIONS:
Device: Placebo PBMT — The PBMT treatments will be performed using the Multi Radiance Medical™ Super Pulsed Laser MR4™console (Solon, OH, USA), with the LS50 (emitter with an area of 20 cm2) and SE25 (emitter with an area of 4 cm2) cluster probes as emitters. Nine sites will be irradiated at patient's lumbar region: 3 central sites, using the SE25 (without any dose, 0 J); and 6 sites in the same direction, but laterally (both sides, 3 at a side), using the LS50 (without any dose, 0 J). Patients will be treated in a single session and they will receive a total dose of 0 J.
  Arms: Placebo PBMT
Device: Active PBMT — The PBMT treatments will be performed using the Multi Radiance Medical™ Super Pulsed Laser MR4™ console (Solon, OH, USA), with the LS50 (emitter with an area of 20 cm2) and SE25 (emitter with an area of 4 cm2) cluster probes as emitters. Nine sites will be irradiated at patient's lumbar region: 3 central sites, using the SE25 (3000 Hz of frequency, 3 minutes of irradiation per site, 24.75 J per site, a totalizing 74.25 J irradiated from SE25); and 6 sites in the same direction, but laterally (both sides, 3 at a side), using the LS50 (1000 Hz of frequency, 3 minutes of irradiation per site, 24.30 J per site, a total of 145.80 J irradiated from LS50). Patients will be treated in a single session and will receive a total dose of 220.05 J.
  Arms: Active PBMT

SUMMARY:
Low back pain (LBP) is ranked as one of the most prevalent health conditions. It is likely that some inflammatory mediators could be associated with pain and disability in these patients. Photobiomodulation therapy (PBMT) is a non-pharmacological therapy often used in patients with LBP that decrease release of inflammatory mediators and accelerate muscle repair in different muscle skeletal conditions, as mechanisms of action. The present research project aims to evaluate the effects of PBMT on systemic levels of inflammatory markers and levels of pain intensity in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
This is a randomized, triple-blinded (therapist, assessor and patient), placebo-controlled trial, with voluntary patients with non-specific chronic low back pain.

Eighteen patients will be randomly allocated to two treatment groups: Placebo or PBMT and one single session of treatment will be provided.

The data will be collected by a blinded assessor and the outcomes of interest it will be levels of inflammatory markers and pain intensity and it will be collected at baseline and 15 minutes after the single session of treatment.

The statistical analysis will follow the intention-to-treat principles. The findings will be tested for their normality using the Shapiro-Wilk test. Parametric data will be expressed as mean and standard deviation and non-parametric data as median and respective upper and lower limits. Parametric data will be analyzed by two-way repeated measures analysis of variance (ANOVA; time versus experimental group) with post-hoc Bonferroni correction. Non-parametric data will be analyzed using the Friedman test and, secondarily, the Wilcoxon signed-rank test.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic non-specific low back pain (defined as pain or discomfort between the costal margins and the inferior gluteal folds, with or without referred symptoms in the lower limbs, for at least 3 month);
* with a pain intensity of at least 3 points measured by a 0-10 points pain numerical rating scale;
* aged between 18 and 65 years;

Exclusion Criteria:

* evidence of nerve root compromise (i.e. one or more of motor, reflex or sensation deficit);
* serious spinal pathology (such as fracture, tumor, inflammatory and infectious diseases);
* serious cardiovascular and metabolic diseases;
* previous back surgery;
* pregnancy.
* severe skin diseases (eg. skin cancer, erysipelas, severe eczema, severe dermatitis, severe psoriasis and severe hives lupus);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Levels of prostaglandin E2 (PGE2) | 15 minutes after the treatment
  Inflammation will be measured by blood samples

SECONDARY OUTCOMES:
Levels of tumor necrosis factor alpha (TNF-a) | 15 minutes after the treatment.
  Inflammation will be measured by blood samples.
Levels of interleukin-6 (IL-6) | 15 minutes after the treatment
  Inflammation will be measured by blood samples
Pain Intensity | 15 minutes after the treatment.
  Pain intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain Numerical Rating Scale), with 0 being "no pain" and 10 "the worst possible pain".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon requested of principal investigator.
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Tomazoni SS, Costa LOP, Joensen J, Stausholm MB, Naterstad IF, Ernberg M, Leal-Junior ECP, Bjordal JM. Photobiomodulation Therapy is Able to Modulate PGE2 Levels in Patients With Chronic Non-Specific Low Back Pain: A Randomized Placebo-Controlled Trial. Lasers Surg Med. 2021 Feb;53(2):236-244. doi: 10.1002/lsm.23255. Epub 2020 Apr 24. PMID 32330315
- [Derived] Tomazoni SS, Costa LOP, Joensen J, Stausholm MB, Naterstad IF, Leal-Junior ECP, Bjordal JM. Effects of photobiomodulation therapy on inflammatory mediators in patients with chronic non-specific low back pain: Protocol for a randomized placebo-controlled trial. Medicine (Baltimore). 2019 Apr;98(15):e15177. doi: 10.1097/MD.0000000000015177. PMID 30985704